CLINICAL TRIAL: NCT02421094
Title: Phase 2 Study to Evaluate Non-Invasive Imaging Methods in Efficacy Assessment of GR-MD-02 for the Treatment of Liver Fibrosis in Patients With NASH With Advanced Fibrosis
Brief Title: Clinical Trial to Evaluate Efficacy of GR-MD-02 for Treatment of Liver Fibrosis in Patients With NASH With Advanced Fibrosis
Acronym: NASH-FX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT-028
Record Dates: First submitted 2015-04-13; First posted 2015-04-20 (Estimated); Results first posted 2020-09-28 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — belapectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GR-MD-02 (Active Comparator): Active
  Interventions: Drug: GR-MD-02
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GR-MD-02 — GM-MD-02 active
  Other Names: galactoarabino-rhamnogalacturonate
  Arms: GR-MD-02
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Controlled, Double-blind, Parallel Group, Single Center Phase 2 Clinical Trial to Evaluate Multiple Non-Invasive Liver Fibrosis Imaging Methods in the Assessment of the Efficacy of GR-MD-02 for the Treatment of Liver Fibrosis in Patients with NASH with Advanced Fibrosis

DETAILED DESCRIPTION:
The primary objective is to determine the difference between placebo and GR-MD-02 treatment in the baseline adjusted mean change in liver fibrosis as measured by corrected T1 (cT1) mapping as determined from LiverMultiScan (LMS), a multi-parametric MRI protocol.

Secondary objectives include evaluating differences between subjects treated with GR-MD-02 versus placebo in:

* The baseline-adjusted change in liver stiffness as measured by MR-elastography
* The baseline-adjusted change in liver stiffness as measured by FibroScan® scores.

An exploratory objective will be to evaluate the correlation of the three diagnostic modalities of LiverMultiScan, MR-Elastography, and FibroScan®.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have liver biopsy demonstrating NASH with Brunt Stage 3 fibrosis within 12 months of randomization. The subject is ≥ 18 years of age and ≤ 75 years old at the time of screening
* The subject is willing and able to provide written informed consent
* The subject is not pregnant and must have a negative pregnancy test prior to start of the study. Post-menopausal women must have been amenorrheic for at least 12 months to be considered of non-child-bearing potential.
* Fertile men and women participating in heterosexual relations must agree to use effective means of contraception throughout their participation in this study and for 90 days after discontinuation of study medication.
* Lactating females must agree to discontinue nursing before the start of study treatment and refrain from nursing until 90 days after discontinuation of study medication.
* Male subjects must refrain from sperm donation throughout the study period and for a period of 90 days following the last dose of study drug.

Exclusion Criteria:

* A history of hepatic decompensation including any episode of variceal bleeding, clinically detectable ascites, or overt hepatic encephalopathy.
* Status post TIPS (Transjugular Intrahepatic Porto-systemic Shunt) procedure.
* Evidence of other forms of chronic liver disease including viral hepatitis B or C, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson's disease, alpha-1 antitrypsin deficiency, alcoholic hepatitis, hemochromatosis, liver cancer, or history of biliary diversion.
* Any of the following laboratory values: Serum alanine aminotransferase (ALT) and aspartate aminotransferase levels > 10X upper limits of normal, Serum creatinine ≥ 2.0 mg/dL, Platelet count < 60,000/mm3, Serum albumin ≤ 2.8 g/dL, INR ≥ 1.7, Direct bilirubin ≥ 2.0 mg/dL
* A MELD score ≥ 15 or Child-Pugh-Turcotte Stage B or C
* Known positivity for Human Immunodeficiency Virus (HIV) infection
* Any subject who had major surgery within 8 weeks of Day 1, significant traumatic injury, or anticipation of need for major surgical procedure during the course of the study.
* Weight reduction surgery within the past 3 years.
* Any subject with current, significant alcohol consumption or a history of significant alcohol consumption for a period of more than 3 consecutive months any time within 1 year prior to screening will be excluded.
* Any subject with concurrent infection including diagnoses of fever of unknown origin (FUO) (subjects must be afebrile at the start of therapy).
* Any history of malignancy, except for the following adequately-treated non metastatic basal cell skin cancer; any other type of skin cancer, except melanoma, that has been adequately treated and has not recurred for at least 1 year prior to enrollment; and adequately treated in situ cervical cancer that has not recurred for at least 1 year prior to enrollment.
* Participation in an investigational new drug (IND) trial in the 30 days before randomization
* Clinically significant medical or psychiatric condition considered a high risk for participation in an investigational study.
* Failure to give informed consent
* Subjects with known allergies to the study drug or any of its excipients.
* Is an employee or family member of the investigator or study site personnel.
* Any subject who cannot undergo an MRI, e.g., due to certain metal or electronic device implants, as determined by the Principal Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- GR-MD-02 8 mg/kg: Active
  GR-MD-02: GM-MD-02 active
Period: Overall Study
Arm/Group | GR-MD-02 8 mg/kg | Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GR-MD-02 8 mg/kg | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (6.19) | 56.7 (6.15) | 58.2 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 13 | 15 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Liver Fibrosis of Corrected T1 (cT1) Mapping (LiverMultiScan -LMS)
Description: Difference in baseline adjusted mean change in liver fibrosis of corrected T1 (cT1) mapping with LiverMultiScan (LMS).
  LiverMultiScan is CE marked as a class IIa medical device. Corrected T1 (cT1) is a Magnetic Resonance (MR) relaxation parameter/measure from the device.The measure cT1 can be compared across different Magnetic Resonance Imaging (MRI) systems and sites. It is an emerging biomarker for rapid quantification of hepatic fibro-inflammatory disease. In unhealthy tissue, such as in inflamed and fibrotic tissues, measures result in longer cT1-relaxation.
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: milliseconds (ms)
Arm/Group | GR-MD-02 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 15
milliseconds (ms) | 19.15 [-7.7 to 43.5] | 1.25 [-7.7 to 43.5]
Statistical Analysis 1: Comparison: GR-MD-02 8 mg/kg vs Placebo; Test type: Superiority; p = 0.1621, ANCOVA

2. Secondary Outcome: Baseline-adjusted Change in Liver Stiffness With MR-elastography (MRE)
Description: Baseline-adjusted change in liver stiffness as measured by MR-elastography. Magnetic resonance elastography (MRE) is a technology that uses MRI imaging with low-frequency vibrations to create a visual map (elastogram) that shows stiffness of body tissues. Currently, MRE is used to detect stiffening of the liver caused by fibrosis and inflammation in chronic liver disease. Liver stiffness increases with liver damage/disease.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Kilopascals, kPa
Arm/Group | GR-MD-02 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 15
Kilopascals, kPa | 0.17 (0.55) | 0.18 (0.63)
Statistical Analysis 1: Comparison: GR-MD-02 8 mg/kg vs Placebo; Test type: Superiority; p = 0.9835, ANCOVA

3. Secondary Outcome: Baseline-adjusted Change in Liver Stiffness by FibroScan®
Description: Baseline-adjusted change in liver stiffness as measured by FibroScan® scores. FibroScan measures scarring by measuring the stiffness of your liver. The fibrosis result is measured in kilopascals (kPa). It's normally between 2 and 6 kPa. Many people with liver disease(s) have a result that's higher than the normal range.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Kilopascals, kPa
Arm/Group | GR-MD-02 8 mg/kg | Placebo
Number analyzed (Participants) | 15 | 15
Kilopascals, kPa | 1.11 (9.51) | -2.32 (5.87)
Statistical Analysis 1: Comparison: GR-MD-02 8 mg/kg vs Placebo; Test type: Superiority; p = 0.2660, ANCOVA

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | GR-MD-02 8 mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/15 | 11/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GR-MD-02 8 mg/kg (N=15) | Placebo (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Food allergy (General disorders) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac murmur (Cardiac disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palmar erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No